CLINICAL TRIAL: NCT03695796
Title: French Cohort for the Study of Non-invasive Tests of Liver Lesions in NAFLD/NASH (FreSH Cohort)
Acronym: FreSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC18_0076
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: NAFLD
Keywords: patients with a NAFLD proven by liver biopsy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: biopsy-proven NAFLD patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): Only one arm because diagnostic study evaluating non-invasive tests using liver biopsy as reference
  Interventions: Diagnostic Test: biopsy-proven NAFLD patients with non-invasive tests of liver fibrosis (blood tests, elastography devices) and biobank

INTERVENTIONS:
Diagnostic Test: biopsy-proven NAFLD patients with non-invasive tests of liver fibrosis (blood tests, elastography devices) and biobank — To evaluate and improve the non-invasive diagnosis of liver fibrosis in NAFLD and to develop the non-invasive diagnosis of NASH

SUMMARY:
Currently, the management of non-alcoholic fatty liver disease (NAFLD) patients has two main limitations. First, there is no approved treatment in NAFLD. Second, liver biopsy remains the reference procedure for the evaluation of liver lesions but it is invasive and can't be proposed to all NAFLD patients who represent 25% of the general population. Phase III trials have recently started in NAFLD with the hope of new treatments available in few years on the market. Consequently, we now need to develop and validate the non-invasive tools that will allow the identification of the subset of NAFLD patients who will benefit from treatment with the new drugs once they will be available in clinical practice.

We aim to generate of large multicenter cohort of biopsy-proven NAFLD patients including non-invasive tests of liver lesions (blood tests, elastography devices) and a biobank to promote a research network in the field of non-invasive diagnosis of liver lesions in NAFLD. Eight French centers highly experienced in this field of research will participate to the cohort.

Our primary aim will be to evaluate and improve the non-invasive diagnosis of liver fibrosis in NAFLD. The primary endpoint will be advanced fibrosis as defined by fibrosis stages F3/4 by the NASH-CRN histological semi-quantitative scoring

ELIGIBILITY:
Inclusion Criteria:

* NAFLD diagnosis defined by the presence of at least two of the following elements:

  * Liver steatosis (hyperechoic liver on hepatic ultrasound, quantification > 5.6 % by spectroscopy or MRI)
  * Presence of one metabolic risk factor:

    * BMI ≥ 25 kg/m2 or waist circumference ≥ 94 cm (male) / ≥ 80 cm (female)
    * Antihypertensive treatment or systolic BP ≥ 130 mmHg or diastolic BP ≥ 85 mmHg
    * Antidiabetic treatment or fasting blood glucose ≥ 5.6 mmol/l
    * Lipid-lowering treatment or triglycerides ≥ 1.71 mmol/l or HDL cholesterol <1.1 mmol/l (male) / <1.3 mmol/l (female)
    * Dysmetabolic hyperferritinemia
  * Anomaly in the liver enzyme test or liver function tests
* Indication for liver biopsy in the clinical management of the patient
* Obtaining the signature of the consent to participate in the study

Exclusion Criteria:

* Steatogenic treatment (corticosteroids, tamoxifen, amiodarone, methotrexate)
* Excessive alcohol consumption in the last 5 years (> 210 g / week for men or > 140 g / week for women)
* Chronic infection with hepatitis B or C
* Any evidence of other concomitant chronic liver disease
* Decompensated cirrhosis (ascites, digestive bleeding due to varicose vein rupture, liver failure, hepatocellular failure, hepato-renal syndrome)
* Hepatocellular carcinoma
* Pregnant, breastfeeding or parturient women
* Persons deprived of their liberty by judicial or administrative decision
* Persons subject to legal protection measures
* Persons unable to consent
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Advanced fibrosis in NAFLD | 1 day
  Advanced fibrosis defined by a stage of fibrosis F≥ 3 on liver biopsy according to the semi-quantitative histological classification of NASH CRN

SECONDARY OUTCOMES:
Non alcoholic steatohepatitis | 1 day
  On liver biopsy (NASH CRN classification): steatosis >=1 AND ballooning >=1 AND lobular inflammation >= 1
Validate the diagnostic performance and thresholds of 2nd generation blood tests compared to 1st generation blood tests | 1 day
Validate the diagnostic performance and thresholds of new elastography devices for the assessment of hepatic fibrosis and steatosis | 1 day
Validate the reliability criteria for Fibroscan in NAFLD, in particular for the XL probe | 1 day
Defining reliability criteria for Acoustic Radiation Force Impulse and Supersonic Shearwave Imaging in NAFLD | 1 day
Validating the performance of the eLIFT algorithm for screening advanced liver fibrosis in NAFLD | 1 day
Assessing the prognostic value of non-invasive fibrosis tests for predicting death from liver-related causes | 1 day
Identify new biomarkers for the non-invasive diagnosis of NASH thanks to collaborations developed by the investigating centres with teams with expertise in 'omics' technologies | 1 day
Estimate the correlation between a new serum marker, phosphatydylethanol, and alcohol consumption in patients with non-alcoholic fatty liver disease | 1 day

CONTACTS AND LOCATIONS:
Locations (16):
- France (15):
  - Amiens University Hospital, Amiens
  - University Hospital of Besançon, Besançon
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - Grenoble University Hospital, Grenoble
  - Hospital of Le Havre, Le Havre
  - University Hospital of Lille, Lille
  - Hospital Center Of Lorient, Lorient
  - Edouard Herriot Hospital, Lyon
  - Saint-Joseph Hospital, Marseille
  - University Hospital Of Nice, Nice
  - University of Bordeaux, Pessac
  - University Hospital of Rouen, Rouen
  - University Hospital of Strasbourd, Strasbourg
  - University Hospital of Toulouse, Toulouse
  - University Hospital Of Nancy, Vandœuvre-lès-Nancy
- University Hospital of Pointe à Pitre, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No